CLINICAL TRIAL: NCT07021768
Title: Controlled, Double-blind, Randomized Clinical Trial of the Use of Laser Auriculotherapy for the Treatment of Low Back Pain
Brief Title: Laser Auriculotherapy for the Treatment of Low Back Pain
Acronym: Laser
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marcelo Neubauer de Paula (Other)
Collaborators: Hospital das Clínicas, University of Sao Paulo Medical School (Unknown)
Responsible Party: Sponsor-Investigator, Marcelo Neubauer de Paula, Guest Professor at the IOTHCFMUSP Acupuncture Center, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 87524325.0.0000.0068
Record Dates: First submitted 2025-05-27; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
Keywords: Laser; Auriculotherapy; Low Back Pain; Nogier; French Auriculotherapy
MeSH Terms: conditions — Low Back Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The procedure will be performed by an unblinded investigator. The patient will be blinded by means of an eye shield that blocks his/her vision. The assessment of pain scales and algometry will be performed by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser auriculotherapy (Experimental): French Laser Auriculotherapy using the ECCO REABILITY device and dual pen with red laser with 660 nm wavelength, both manufactured by Ecco Optical Fibers and Devices, using the ideal Nogier Frequency for each region with application of 2 J per point with 100 mW power. For the active group, a 120 mW active tip, red laser with 660 nm, pulse width of 1.2 milliseconds will be used.
  Interventions: Device: Laser Auriculotherapy
- Placebo auriculotherapy (Placebo Comparator): Placebo laser through the ECCO REABILITY device and sham pen both manufactured by Ecco Optical Fibers and Devices. For the control group, a placebo tip with a 660 nm red laser with 1 mW of power and a pulse width of 1.2 milliseconds will be used.
  Interventions: Device: Laser Auriculotherapy

INTERVENTIONS:
Device: Laser Auriculotherapy — French Laser Auriculotherapy using the ECCO REABILITY device and dual pen with red laser with 660 nm wavelength, both manufactured by Ecco Optical Fibers and Devices, using the ideal Nogier Frequency for each region with application of 2 J per point with 100 mW power. For the active group, a 120 mW active tip, red laser with 660 nm, pulse width of 1.2 milliseconds will be used.
  Other Names: Photobiomodulation

SUMMARY:
Controlled, double-blind, randomized clinical trial

Primary endpoint:

To demonstrate the superiority of Laser French Auriculotherapy (AFL) in relieving pain in patients with low back pain after a single session.

Primary outcome:

The increase in pain tolerance will be assessed by Algometry of the affected muscles

Secondary endpoints:

To determine the duration of the analgesic effect of AFL. To determine the increase in pain tolerance through Algometry

Secondary outcomes:

The improvement in pain after treatment with daily measurements for 7 days will be assessed using the TotPar Scale The reduction in pain will be assessed using the Sum of Pain Intensity Difference (SPID) Scale by comparing the differences in scores observed between pre-treatment and post-treatment with daily measurements for 7 days Reduction in the 10-point visual analogue scale for pain. Need for rescue medication

Safety endpoint:

Evaluate adverse events that occurred during the trial, after signing the Informed Consent Form (ICF).

Safety outcomes:

Evaluate safety through data obtained in clinical and physical assessments, and in specific assessments of the clinical trial (immediately after signing the ICF).

Evaluate the rate of occurrence of non-serious and serious adverse events, related and unrelated to the treatment groups throughout the clinical trial.

DETAILED DESCRIPTION:
Trial Population Patients with primary or secondary low back pain, aged between 18 and 65 years, who attended the Institute of Orthopedics and Traumatology of the Hospital das Clínicas of the Faculty of Medicine of the University of São Paulo (IOTHCFMUSP) acupuncture clinic.

Trial Design

Clinical, superiority, double-blind, randomized trial with two parallel groups:

* Test Group: Will receive an auricular laser application at the points indicated for this treatment and that are active (through a point locator device) using a 660 nanometer red laser with the appropriate Nogier frequency, 2 joules per point. In addition, an infrared laser will be applied at the frequency
* Comparator group: will receive a touch on the skin at the same points with a non-laser emitting pen.

Both patients will wear opaque protective glasses and, therefore, will not be able to observe the application. The patient must continue to use the prescribed medications.

Experimental procedure:

Laser French Auriculotherapy using the ECCO REABILITY device and dual pen with red laser with a wavelength of 660 nm, manufactured by Ecco Fiber Optics and Devices, using the ideal Nogier Frequency for each region, with the application of 2 J per point and a power of 100 mW. For the active group, a 120 mW active tip, red laser with 660 nm, pulse width of 1.2 milliseconds will be used.

Comparator procedure:

Placebo laser using the ECCO REABILITY device and sham pen, both manufactured by Ecco Fiber Optics and Devices. For the control group, a placebo tip with red laser 660 nm with 1 mW of power, pulse width of 1.2 milliseconds will be used.

Application method Single session. The auriculotherapy treatment protocol will be adapted according to each patient. The Nogier mapping will be applied: lumbar and sacral spine area; Lumbar muscles in the posterior wall, thalamus, zero, zero', Shen Men and prefrontal cortex, main sensory and master point of the spine, in addition to the radian technique using the corresponding point in the auricular helix. The points to be used must be active according to the EL30 Finder differential pen point locator device manufactured by NKL Medical DevicesL.

A red laser with a wavelength of 660 nm will be used with the ideal frequency for each location (Nogier frequencies) with an intensity of 2 joules per point. Patients randomized to the placebo group will undergo the same procedures, however a placebo pen will be used.

If the pain is located on one side, the application will be made in the ear on the same side as the affected side. If the pain is bilateral, the application will be made in both ears. If the pain only affects the midline, the application will be made in the ear on the same side as the dominant hand.

Methodology Blinding The procedure will be performed by an unblinded investigator. The patient will be blinded by means of an eye protector that blocks his/her vision. The assessment of pain scales and algometry will be performed by a blinded investigator.

There will be 11 visits in total Visit 0 (V0) - Initial visit

* Participant clarification about the protocol
* Signing of the informed consent form
* Assessment of the inclusion and exclusion criteria;
* Randomization of the research participant; This visit will be performed by an unblinded investigator

Visit 1 (V1) - Screening visit

After the participant consents to participate in the trial, the following procedures must be performed:

* Collect demographic data;
* Assess and record medical history;
* Perform a complete physical examination;
* Record previous medications used in the last two weeks;
* Apply the initial scales
* Test algometry on the muscles affected by pain. This visit will be performed by a blinded investigator

Visit 2 (V2) - Randomization and treatment visit • Apply the experimental or sham treatment according to randomization This visit will be performed by an unblinded investigator

Visit 3 (V3) - Reassessment visit

• Reapply the TotPar and SPID scale and repeat algometry This visit will be performed by a blinded investigator

Visit 4 (V4) - Telephone reassessment visit

* After 24h of V3
* Reapply the TotPar and SPID scale This visit will be performed by a blinded investigator

Visit 5 (V5) - Telephone reassessment visit

* After 24h of V4
* Reapply the TotPar and SPID scale This visit will be performed by a blinded investigator

Visit 6 (V6) - Telephone reassessment visit

* After 24h of V5
* Reapply the TotPar and SPID scale SPID This visit will be conducted by a blinded investigator

Visit 7 (V7) - Telephone reassessment visit

* After 24h from V6
* Reapply the TotPar and SPID scale This visit will be conducted by a blinded investigator

Visit 8 (V8) - Telephone reassessment visit

* After 24h from V7
* Reapply the TotPar and SPID scale This visit will be conducted by a blinded investigator

Visit 9 (V9) - Telephone reassessment visit

* After 24h from V8
* Reapply the TotPar and SPID scale This visit will be conducted by a blinded investigator

Visit 10 (V10) - Closing visit

* After 24h from V9
* Reapply the TotPar and SPID scale
* Final reassessment
* Referral for follow-up This visit will be conducted by a blinded investigator.

Statistical Plan The outcome is of an ordinal qualitative nature and, therefore, the one-tailed non-parametric Mann-Whitney-Wilcoxon test will be used to verify whether laser is superior to sham acupuncture in reducing pain.

The outcome is of an ordinal qualitative nature and, therefore, the Fischer test will be used to verify whether laser is superior to sham acupuncture in reducing pain. The sample size calculation was performed using the G*Power software, considering that the statistical analysis will be performed using the Fisher test:

* Fisher's Exact Test
* One-tailed Hypothesis Test
* Two independent groups
* Options: Exact distribution
* Input: Tail(s) = One
* Proportion p1 = 0.8
* Proportion p2 = 0.5
* Significance Level (α error) = 0.05
* Power (1-β error) = 0.95
* Allocation ratio N2/N1 = 1
* Output: Sample size group Active Laser Group = 59
* Sample size group Placebo Group = 59
* Total sample size = 118
* Real power = 0.9521908
* Real α = 0.0399172 Randomization will be stratified by gender and the sequence will be generated by the SEALED ENVELOPE portal available at https://www.sealedenvelope.com/.

Blinding The study will be double-blind, with the participation of a blinded investigator and an unblinded investigator.

Source of Patients for the study Patients who were referred to the outpatient clinic of the Acupuncture Center of the IOTHCFMUSP.

ELIGIBILITY:
Inclusion Criteria:

* Participant capable of understanding and performing all procedures and instructions described in the Informed Consent Form approved by the Research Ethics Committee;
* Participants of both sexes, aged between 18 and 65 years (inclusive);
* Participants diagnosed with low back pain who are in pain at the time of the assessment

Exclusion Criteria:

* Any clinical observation finding (clinical/physical evaluation) that is interpreted by the investigating physician as a risk to participation in the clinical trial;
* Patient with a deforming lesion on the ear
* Patient with a tattoo covering any of the points selected for treatment
* Patients using ear expanders on the side to be treated
* Research participants who have participated in clinical trial protocols in the last 12 (twelve) months (Brazilian National Health Council Resolution 251, of August 7, 1997), unless the investigator believes that there may be direct benefit to the same.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Algometry | 1 hour after intervention
  Increase in pain tolerance will be assessed by Algometry of the affected muscles

SECONDARY OUTCOMES:
TotPar Scale | 1 week after intervention
  The improvement in pain after treatment with daily measurements for 7 days will be assessed using the TotPar Scale.
SPID Scale | 1 week after intervention
  The reduction in pain will be assessed using the SPID Scale by comparing the differences in scores observed between pre-treatment and post-treatment with daily measurements for 7 days.
Visual analogue scale | 1 week after intervention
  Reduction in the 10-point visual analogue scale for pain.
Rescue medication | 1 week after intervention
  Need for rescue medication
Adverse Events | 1 week after intervention
  Assess the rate of occurrence of non-serious and serious adverse events, related and unrelated to the treatment groups, throughout the clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo N de Paula, PHD Student, Principal Investigator — Faculty of Medicine of the University of São Paulo; Wu T Hsing, PHD, Study Chair — Faculty of Medicine of the University of São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Initially the data will be anonymized and will be available for possible auditing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For 12 months after the study is published
Access Criteria: Members of the board of the journal to which the study was submitted, members of the doctoral defense committee, research ethics committee, members of the board of directors of the institution where the study will be carried out